CLINICAL TRIAL: NCT01526798
Title: Improvement of EPO-resistance in HD Patients With Chronic Inflammation by High Cut-off Hemodialysis - Pilot Study (CIEPO-PILOT)
Brief Title: Improvement of EPO-resistance in Hemodialysis Patients With Chronic Inflammation by High Cut-off Hemodialysis
Acronym: CIEPO-PILOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Dialysatoren GmbH (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No 1491 CIEPO-PILOT
Record Dates: First submitted 2012-02-02; First posted 2012-02-06 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: End-Stage Renal Disease (ESRD)
Keywords: End-Stage Renal Disease (ESRD); chronic Inflammation; EPO Resistance; ESA Resistance; high cut-off dialysis; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therlite hemodialysis (Experimental)
  Interventions: Device: Theralite (high cut-off hemodialysis)
- Control group hfHDF (Active Comparator): Control group hfHDF
  Interventions: Device: Conventional high-flux dialyzer

INTERVENTIONS:
Device: Theralite (high cut-off hemodialysis) — Hemodialysis with Theralite dialyzer alternating with standard high-flux dialyzer
  Arms: Therlite hemodialysis
Device: Conventional high-flux dialyzer
  Arms: Control group hfHDF

SUMMARY:
Chronic inflammation in dialysis patients is linked to cardiovascular mortality and clinical signs and symptoms, like the impaired response to erythropoiesis-stimulating agents (ESAs). This study aims to demonstrate that high cut-off hemodialysis is effective in reducing chronic inflammation and thereby improving response to ESAs.

DETAILED DESCRIPTION:
Chronic inflammation in hemodialysis patients (micro-inflammation) is caused by multiple inflammatory stimuli and becomes apparent by elevated levels of biochemical markers such as CRP, IL-6, cellular activation markers etc. Chronic inflammation is linked to clinical signs and symptoms and cardiovascular mortality in dialysis patients. Inflamed dialysis patients show impaired response to erythropoiesis-stimulating agents (ESA) related to reduced iron utilization (functional iron deficiency) and elevated CRP levels are associated with a greater need for ESA to meet hemoglobin targets. If absolute iron deficiency can been excluded, EPO resistance is likely related to 'inflammatory block'.

The high molecular permeability of the Theralite high cut-off membrane allows for significant clearance of cytokines and other pro-inflammatory solutes by hemodialysis as shown in previous trials with high cut-off dialyzers. The study therefore aims to demonstrate that Theralite dialysis is effective in reducing chronic inflammation in ESRD patients, thereby improving EPO responsiveness. If this can be demonstrated, application of Theralite hemodialysis may reduce morbidity and mortality in the long term in ESRD patients.

ELIGIBILITY:
Inclusion Criteria:

* ESRD treated with chronic HD for at least 3 months
* Treatment with high-flux dialyzers for at least 3 months
* Age ≥18 years
* Receiving ESA to treat anemia for at least 3 months
* Impaired ESA responsiveness as indicated by EPO resistance index > median of patients in study center
* Transferrin saturation (TSAT) ≥20% (last routine value prior to randomization)
* Serum ferritin ≥100 ng/ml (last routine value prior to randomization)

Exclusion Criteria:

* Acute infection ≤4 weeks prior to randomization
* HIV or hepatitis infection
* Catheter
* Chronic liver disease
* Active cancer
* Known blood dyscrasia (paraprotein abnormalities)
* Known bleeding disorders
* Bleeding episode ≤12 weeks prior to randomization
* Blood/red cell transfusion ≤12 weeks prior to randomization
* Hypoalbuminemia defined as serum albumin concentration below 35 g/L (last routine value prior to randomization)
* Participation in another clinical interventional investigation
* Pregnancy
* Inability to give informed consent
* Planned transplantation within study period +3 months
* Planned interventions requiring hospitalization >1 week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Erythropoietin (EPO) resistance index | 12 weeks after randomization
  Weekly EPO dose in international units (IU) per kg body weight divided by hemoglobin value in g/dL

SECONDARY OUTCOMES:
high sensitivity C-reactive protein (CRP), hepcidin, Free Light Chains (FLC), Interleukin (IL)-6, Interleukin (IL)-10 | baseline, 4, 8 and 12 weeks
  Change in pre-dialysis concentration over study period
Urea, Hepcidin, Free Light Chains, IL-6, IL-10 | baseline, week 1
  Pre- and post-dialysis concentration of urea, hepcidin
Albumin | baseline, weeks 2,4,6,8,10,12,14,16,18,20,22,24
  Pre-dialysis albumin concentration during study period and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Teatini, Dr., Principal Investigator — Azienda Ospedaliera Garbagnate Milanese Ospedale Bollate - Divisione Nefrologia e Dialisi
Locations (1):
- Azienda Ospedaliera Garbagnate Milanese Ospedale Bollate - Divisione Nefrologia e Dialisi, Bollate, Milan, Italy